CLINICAL TRIAL: NCT02621346
Title: Maintaining Muscle Mass Gains
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Alison Divine, PhD Candidate, Western University, Canada
Allocation: Randomized | Model: Factorial | Masking: Single
Other Study IDs: HSREB 107286
Record Dates: First submitted 2015-12-01; First posted 2015-12-03 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Using Imagery to Maintain Muscle Mass Gains in the Quadriceps

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Imagery Group (Experimental): The imagery group, will sit on the leg press and image completing 3 sets of leg press. The imagery group will be asked to fill out the Movement Imagery Questionnaire -revised as this gives us a measure of imagery ability. The imagery group will be given an imagery script prior to imaging. Weekly manipulation checks will be completed to ensure that participants are imagining what they are supposed to.
  Interventions: Behavioral: Imagery
- Maintenance Group (Active Comparator): The maintenance group will continue to perform the leg press three times per week at 1/3rd of final strength assessment. This is the percentage of intensity recommended to maintain muscle mass and strength gains by the American College of Sports Medicine.
  Interventions: Behavioral: Muscle Maintenance
- Control Group (Active Comparator): Control group will come in 3 times per week for 20 minutes and complete 3 sets of 8-12 of a bicep curl 1/3 of predicted 1 RM
  Interventions: Behavioral: Bicep Curls

INTERVENTIONS:
Behavioral: Imagery — Prior to exercising participants will be given an imagery script. Afterwards, participants will imagine completing the leg press.
  Arms: Imagery Group
Behavioral: Muscle Maintenance — Participants complete the leg press exercises at an intensity that promotes muscle maintenance but not muscle growth
  Arms: Maintenance Group
Behavioral: Bicep Curls — Control group participants will complete a bicep exercise at a maintenance training intensity.
  Arms: Control Group

SUMMARY:
Mental imagery is effective for improving motor skills as well as increasing muscles strength and size. Strength is also maintained after immobilization of a muscles when engaging in imagery. This may have important implications for rehabilitation settings and for sedentary individuals. We may not be able to get people wot exercise but if they can maintain muscles size and strength via imagery this may have beneficial health and functional outcomes.

DETAILED DESCRIPTION:
It is well established that imagery improves motor performance and learning. Imagery is defined as "an experiences that mimics real experiences, and involves using a combination of different sensory modalities in the absence of actual perception: (Cumming & Ramsey, 2009, p.5). The mechanism thought to enhance the effectiveness of imagery is through the theory of functional equivalence (Holmes & Collins, 2001). This theory proposes that when a person images, they activate similar areas of the brain, which also become active if the individual actually engages in the task. The PETTLEP model (Holmes & Collins, 2001) is a framework for the application of the theory of functional equivalence. It is proposed that incorporating each PETTLEP elements into the Imagery experience will increase the similar areas of brain activation and enhance imagery's effectiveness. The elements of the PETTLEP model are as following: 1) physical refers to recreating the physical components of the skill; 2) environment, refers to recreating the place where the skill is performed; 3) task, refers to the specificity of the content of the imagery to the skill being imaged 4) Timing refers to the speed at which imagery is completed. Real times is the most effective; 5) Learning, refers to adapting imagery in response to learning; 6) Emotion refers to the inclusion of related emotions in imagery as this lead to a more real-life situation and enhances the effectiveness of imagery; and 7) perspective refers to the viewpoint through which imagery is done (Holmes & Collins, 2001). With respect to perspective there are three types of views and image can involves. The first is internal perspective, which refers to creating an image of what the individual would see if looking through their eyes. Second is external perspective, which refers to imaging yourself from the outside, as if you were watching yourself in a video. Lastly, is the kinaesthetic perspective, which refers to imaging how the movement feels. Research has shown that for increasing muscles strength and size the internal imagery perspective is more effective than external (Leban et al., 2010; Yoa et al., 2013). Additionally, internal imagery increasing physiological responses, such as hear rate, blood pressure, respiratory rate compared to external imagery (Ranganthen et al., 2004). Research examining the effects of motor imagery on increasing strength has found that imagery is effective. Significant increased in muscles strength have occurred ranging from 10-22% strength increases as a result of imagery (Clark et al., 2014; Leban et al., 2013; Yao et al., 2013). Additionally, research has found effects trending on significant on muscle size (Leban, 2013). Leban and colleagues (2013) trained participants over a total of 12 days, as saw increased in muscles size. Physiological research suggests that the development of muscle mass and size requires 4-8 weeks (American College of Sports Medicine, 2012). As such, given that trending significance was found for the exercise plus imagery group in size of the thigh muscles after a short 12-day training protocol and no difference in size for the exercise only group, this suggests that imagery may affect muscle hypertrophy. Additionally, research has looked at the use of imagery to maintain muscles strength after immobilization. For instance, after immobilization of the index finger, the mental imagery group maintained strength despite muscles atrophy (Yao et al., 1996). Given these findings it is possible that following muscle hypertrophy and strength gains through exercise, imagery may help to attenuate the loss of muscle strength and size in a maintenance phase. This may have importance implications for rehabilitation settings, as well as influences how sedentarianism is approached. For some untrained sedentary individuals, using mental imagery is far easier that exercising. If imagery not only attenuates the loss of strength and muscles size this may help individuals who are not able to exercise maintain their muscles and strength required for functional daily activities. Therefore the purpose of this study is to assess how mental imagery attenuates muscles size and strength over four weeks after an eight-week training program designed to increase muscles hypertrophy and strength. It is hypothesized that the imagery group will maintain their size and strength gains at a similar rate as the maintenance exercise group, whereas the control group is expected to lose muscle gains.

The study consists of two phases. Phase 1 is the exercise phase. Phase 2 is the maintenance phase. The study will be a single blind randomized control trial. PHASE 1: Consenting participants will complete the Par Q health screening, the Godin-Leisure Time Exercise Questionnaire (GLTEQ; Godin & Sheppard, 1985) and a demographic questionnaire. Following this, participants will be given a DEXA body scan to assess muscle mass and a predicted 1rep maximum (1RM) strength test on the leg press. The predicted 1 RM is a submaximal strength test used to estimate the maximum amount of weight an individual can move once. Participants will come into the lab 3 times per week and following a 5 minute walking warm up at 40-60% of the predicted heart rate reserve, will complete 2 warm up leg press sets followed by 3 work sets of 8-12 reps with 1 minute rest between sets. Following this participants will complete 3-5 minute cool down. Each session will last approximately 20 minutes. Participants will start at 70% of and predicted 1RM will increase progressively. A 10%increase in load will be applied when the individual can perform the current workload and 1-2 reps over the required number in the third set. Participants will complete 8weeks of leg press exercises. After 8 weeks participants will be given a DEXA scan and a predicted 1 RM test. For those participants that show muscle growth in the leg muscles on the DEXA will move onto phase 2. PHASE 2: participants that move on to phase 2 will be randomized into 1 of 3 groups. This phase will last for 4 weeks. All three groups will continue to come into the lab three times per week for20 minutes per session. The maintenance group will continue to perform the leg press at 1/3rd of final strength assessment. This is the percentage of intensity recommended to maintain muscle mass and strength gains by the American College of Sports Medicine. The imagery group, will sit on the leg press and image completing 3 sets of leg press. The imagery group will be asked to fill out the Movement Imagery Questionnaire -revised as this gives us a measure of imagery ability. The imagery group will be given an imagery script prior to imaging. Weekly manipulation checks will be completed to ensure that participants are imagining what they are supposed to. Control group will come in 3 times per week and complete 3 sets of 8-12 of a bicep curl 1/3 of predicted 1 RM. Once per week imagery and control participants will be hooked up to EMG to see if there is muscle activation during imagery. The EMG will be placed on surface of the skin of the quadriceps muscles. EMG will be on for the duration of the 15 minutes during the executing of imagery leg presses or the control group bicep curl exercises. The EMG is measured in microvolts. Measuring the above parameter will involve connecting the participants to sensors and electrodes that will pick up on muscle tension responses. This process is non-invasive. Sensors are placed on the surface of the skin. Following the 4 weeks participants will be given another DEXA scan and predicted 1 rep max. At the end of PHASE 2 participants will complete a final predicted 1 RM strength assessment as well as a DEXA scan to measure muscles mass. Additionally, all groups will be given an imagery manipulation check to see if the control or maintenance group imaged during PHASE2.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 of 35. Inclusion criteria is untrained individuals (no history of weight or cardio training) and free of physical disease or orthopedic limitations.

Exclusion Criteria:

* Exclusion criteria includes cognitive impairment leading to the inability to image, orthopaedic illness or injury that prevents engaging in leg exercises and pregnant women due to the radiation rom the DEXA scan.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Muslce mass (grams) determined by the DEXA body scan. | 4 weeks

SECONDARY OUTCOMES:
Muscle strength | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise and health Psychology Lab, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will provided to each participant at the end of the study.

REFERENCES:
- [Background] Clark BC, Mahato NK, Nakazawa M, Law TD, Thomas JS. The power of the mind: the cortex as a critical determinant of muscle strength/weakness. J Neurophysiol. 2014 Dec 15;112(12):3219-26. doi: 10.1152/jn.00386.2014. Epub 2014 Oct 1. PMID 25274345
- [Background] Cumming, J., & Ramsey, R. (2009). Imagery interventions in sport. In S.D Mellalieu & S. Hanton (Eds.)., Advances in applied sport psychology: A review (pp.5-36). London: Routledge
- [Background] Holmes, P. S., & Collins, D. J. (2001). The PETTLEP approach to motor imagery: A functional equivalence model for sport psychologists. Journal of Applied Sport Psychology, 13, 60-83.
- [Background] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Background] Lebon F, Collet C, Guillot A. Benefits of motor imagery training on muscle strength. J Strength Cond Res. 2010 Jun;24(6):1680-7. doi: 10.1519/JSC.0b013e3181d8e936. PMID 20508474
- [Background] Ranganathan VK, Siemionow V, Liu JZ, Sahgal V, Yue GH. From mental power to muscle power--gaining strength by using the mind. Neuropsychologia. 2004;42(7):944-56. doi: 10.1016/j.neuropsychologia.2003.11.018. PMID 14998709
- [Background] Yao, G. H., Wilson, S. L., Cole, K.J., Darline, W.G., Tuh, W. T. C. (1996). Imagined muscle contraction training increases voluntary neural drive to muscle. Journal of Pscyhophysiology, 10, 198-208.
- [Background] Yao WX, Ranganathan VK, Allexandre D, Siemionow V, Yue GH. Kinesthetic imagery training of forceful muscle contractions increases brain signal and muscle strength. Front Hum Neurosci. 2013 Sep 26;7:561. doi: 10.3389/fnhum.2013.00561. eCollection 2013. PMID 24133427